CLINICAL TRIAL: NCT00303030
Title: A Randomized, Controlled, Clinical Trial of Biofeedback and Anal Injections as First Treatment of Fecal Incontinence.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Biofeedback or injections
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Fecal Incontinence
Keywords: Fecal incontinence; Biofeedback; Patient Satisfaction; Quality of LifeTreatment Outcome; Injections
MeSH Terms: conditions — Fecal Incontinence; Patient Satisfaction | interventions — dextranomer-hyaluronic acid copolymer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Anal injection (Active Comparator)
  Interventions: Procedure: 1. Anal injection
- 2. Biofeedback (Active Comparator)
  Interventions: Procedure: 2. Biofeedback

INTERVENTIONS:
Procedure: 1. Anal injection — Submucosal injection just above the linea dentata in the anal canal of 4 x 1 ml of dextranomere.
  Other Names: Solesta
  Arms: 1. Anal injection
Procedure: 2. Biofeedback — Training under the guidance of a physiotherapist with the help of a biofeedback device with an anal probe.
  Arms: 2. Biofeedback

SUMMARY:
A short presentation of a randomized clinical trial of biofeedback and anal injections as a first treatment option of faecal incontinence.

Background: Faecal incontinence affects mainly women who have suffered sphincter disruption from vaginal delivery, but individuals of all ages can be affected. The treatment of this debility is not uniform between institutions or internationally. Often is surgical reconstruction of the anal sphincter performed, or other invasive, costly treatment options.

The study: We intend to conduct a randomized, controlled, clinical trial where we compare the effect of two less invasive, less costly treatment options as a first alternative: biofeedback and anal injections. Our hypothesis is that anal injections will give a better and more lasting effect than biofeedback. The primary endpoint will be change in faecal incontinence assessed by the St. Marks incontinence score. Secondary endpoints will include change in quality of life and several physiological parameters. We intend to include 62 patients in both groups, 124 all together, from 2 centres in Norway. The observation time is 2 years. We plan to include the first patient April 2006, and conclude the study by December 2010. This study can contribute to a more appropriate treatment-algorithm for these patients.

Study group:

* Barthold Vonen MD PhD, Department of gastroenterological surgery, University Hospital of North Norway
* Rolv-Ole Lindsetmo MD PhD, Department of gastroenterological surgery, University Hospital of North Norway
* Arvid Stordahl MD PhD., Department of Surgery, Østfold Hospital Fredrikstad
* Ylva Sahlin MD PhD, Department of Surgery, Innlandet Hospital Hamar
* Trond Dehli, MD, Department of gastroenterological surgery, University Hospital of North Norway
* Kjersti Mevik, Stud. Med, University of Tromso

Project manager: Trond Dehli

Funding, approvals, publication: This study is funded from Northern Norway Regional Health Authority and The Institution of Norwegian Health- and rehabilitation-organizations. It has been approved by the Regional Committee for Medical Research Ethics and Norwegian Social Science Data Services. The results will be published in an international peer-reviewed journal after the Vancouver-convention's guidelines. The results will also be presented at national and international conferences.

Contact:

Trond Dehli, Department of gastroenterological surgery, University hospital North Norway, Breivika, 9038 Tromsø trond.dehli@unn.no tlf: +47 776 26 000

ELIGIBILITY:
Inclusion Criteria:

* Fecal incontinence lasting more than 6 months
* St. Marks score of 4 or more
* No known local or general neurological disease
* 18 years or older
* No constipation

Exclusion Criteria:

* Total rupture of the sphincter of more than 120 degrees
* Diabetes mellitus with late complications (neurological og cardiovascular)
* Ulcus simplex/rectal ulcus
* Anal/rectal prolapse
* ileo-anal anastomosis
* Cancer recti or cancer ani last 2 years
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2006-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Incontinence measured by St.Marks incontinence score | 2 years

SECONDARY OUTCOMES:
Health related Quality of Life measures | 2 years
Physiologic measures | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Barthold Vonen, M.D., Ph.D., Study Director — University of Tromsø, Norway
Locations (3):
- Norway (3):
  - Innlandssykehuset Hamar, Hamar
  - Anorektallaboratoriet, Østfoldsykehuset Sarpsborg, Sarpsborg
  - Avdeling for gastroenterologisk kirurgi, University hospital of North Norway, Tromsø